CLINICAL TRIAL: NCT00001137
Title: Adult AIDS Clinical Trials Group Longitudinal Linked Randomized Trials (ALLRT) Protocol
Brief Title: Long-Term Data Collection From Participants in Adult AIDS Clinical Trials
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5001; 1U01AI068636 (NIH); AACTG A5001
Record Dates: First submitted 2000-01-28; First posted 2001-08-31 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Treatment Naive; Virus Replication; AIDS-Related Opportunistic Infections; HIV-1; Risk Factors; Incidence; RNA, Viral; Anti-HIV Agents; Viral Load; Lipodystrophy; Nervous System; Cardiovascular System; Neurologic Symptoms
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Lipodystrophy; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine what combinations of anti-HIV drugs work best in patients treated over several years. The study will also assess the occurrence of side effects and opportunistic infections in patients with low viral loads compared to those with higher viral loads.

DETAILED DESCRIPTION:
A compilation of outcomes of various antiretroviral therapies would be beneficial when evaluating which strategies are most effective in long-term treatment of HIV-1. Using data from present and recently completed studies, this study will collect information on therapies and their control of HIV infection and maintenance of durable suppression of HIV-1 replication.

No treatment is provided by this study, but patients will continue to receive highly active antiretroviral therapy (HAART) from other studies in which they are coenrolled. Blood and urine collection will occur at study entry and periodically throughout the study. Women may undergo pelvic exams and Pap smears. Portions of blood samples will be stored to evaluate genotypic/phenotypic susceptibility testing. Medical histories, physical exams, and questionnaires will be completed periodically.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 infected
* Enrolled in an AIDS Clinical Trial Group (ACTG) parent study and has enrolled in this study on or before the Week 16 visit of the parent study, including the visit window of the parent study. More information on this criterion can be found in the protocol.
* Willing to provide consent for the release and use of clinical data from the parent study
* Life expectancy of at least 24 weeks
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria

* Active alcohol or drug abuse that may interfere with the study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study will be HIV-infected men and women who are enrolled in an ACTG parent study and are receiving HAART.
Sampling Method: Non-Probability Sample
Enrollment: 5982 (Actual)
Dates: Start 2000-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Successive suppressed viral load measures | Measured 144 weeks after randomization
Genotypic or phenotypic resistance | Measured at baseline and study completion
Complications of HIV disease, including survival, HIV-related opportunistic infections, HIV-related non-opportunistic complications, adverse effects of antiretroviral therapies of grade three or greater | Measured throughout
Absolute number and percentage of CD4 and CD8 T cells | Measured 144 weeks after randomization
Absolute number and percentage of naive cells, including CD4, CD45RA, and CD62L cells | Measured 144 weeks after randomization
Absolute number and percentage of memory cells, including CD4, CD45RO+, and CD45RA- cells | Measured 144 weeks after randomization
Levels of immune activation markers, including CD8, CD38, and HLA-DR cells | Measured 144 weeks after randomization

SECONDARY OUTCOMES:
HIV-1 latency or replication in tissue or cellular reservoirs | Measured at baseline, Week 16, Week 48, and study completion
Syncytium and non-syncytium inducing (SI/NSI) phenotype | Measured at baseline, Week 16, Week 48, and study completion
Metabolic and neurologic complications | Measured at baseline, Week 16, Week 48, and study completion
Immune responses to antigens such as cytomegalovirus (CMV), Myobacterium avium complex (MAC), Candida, and HIV | Measured 144 weeks after randomization
Plasma concentrations of antiretroviral medications other than nucleoside/tide reverse transcriptase inhibitors (NRTIs) | Measured at baseline, Week 16, and study completion
Effect of gender, use of hormonal therapies, presence or absence of menopause on short- and long-term virologic suppression, and pap smear abnormalities | Measured at baseline, Week 48, and study completion
Quality of life scores | Measured at baseline, Week 48, and study completion
Subject-reported patterns of adherence | Measured at baseline, Week 48, and study completion
Estimated inpatient, outpatient, and total costs | Measured at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Constance A. Benson, MD, Study Chair — Division of Infectious Disease, Antiviral Research Center, University of California, San Diego; Ann C. Collier, MD, Study Chair — University of Washington
Locations (77):
- United States (75):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente LAMC, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - UC Davis Med Ctr, Sacramento, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Univ of California, San Francisco/San Francisco General Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - Marin County Specialty Clinic, San Rafael, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Denver Public Health CRS, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Emory Hemo Comp Evaluation Clinic / East TN Comp Hemo Ctr, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Tripler Army Med Ctr, Tripler AMC, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Tulane Med Ctr Hosp, New Orleans, Louisiana
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Wayne State Univ. CRS, Detroit, Michigan
  - Hennepin County Medical Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - AIDS Care CRS, Rochester, New York
  - Community Health Network Inc, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Wake County Department of Health, Chapel Hill, North Carolina
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Presbyterian Medical Center - Univ. of PA, Norristown, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Peabody Health Center CRS, Dallas, Texas
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
  - Univ of Washington, Seattle, Washington
- Puerto Rico (2):
  - Puerto Rico-AIDS CRS, San Juan
  - Univ of Puerto Rico, San Juan

REFERENCES:
- [Background] Jain R, Clark NM, Diaz-Linares M, Grim SA. Limitations of current antiretroviral agents and opportunities for development. Curr Pharm Des. 2006;12(9):1065-74. doi: 10.2174/138161206776055813. PMID 16515486
- [Background] Torre D, Speranza F, Martegani R. Impact of highly active antiretroviral therapy on organ-specific manifestations of HIV-1 infection. HIV Med. 2005 Mar;6(2):66-78. doi: 10.1111/j.1468-1293.2005.00268.x. PMID 15807712
- [Derived] Siddiqui M, Moore TJ, Long DM, Burkholder GA, Willig A, Wyatt C, Heath S, Muntner P, Overton ET. Risk Factors for Incident Hypertension Within 1 Year of Initiating Antiretroviral Therapy Among People with HIV. AIDS Res Hum Retroviruses. 2022 Sep;38(9):735-742. doi: 10.1089/AID.2021.0213. Epub 2022 Aug 23. PMID 35778856
- [Derived] Angelidou K, Hunt PW, Landay AL, Wilson CC, Rodriguez B, Deeks SG, Bosch RJ, Lederman MM. Changes in Inflammation but Not in T-Cell Activation Precede Non-AIDS-Defining Events in a Case-Control Study of Patients on Long-term Antiretroviral Therapy. J Infect Dis. 2018 Jun 20;218(2):239-248. doi: 10.1093/infdis/jix666. PMID 29309629
- [Derived] Coban H, Robertson K, Smurzynski M, Krishnan S, Wu K, Bosch RJ, Collier AC, Ellis RJ. Impact of aging on neurocognitive performance in previously antiretroviral-naive HIV-infected individuals on their first suppressive regimen. AIDS. 2017 Jul 17;31(11):1565-1571. doi: 10.1097/QAD.0000000000001523. PMID 28471765
- [Derived] Riddler SA, Aga E, Bosch RJ, Bastow B, Bedison M, Vagratian D, Vaida F, Eron JJ, Gandhi RT, Mellors JW; ACTG A5276s Protocol Team. Continued Slow Decay of the Residual Plasma Viremia Level in HIV-1-Infected Adults Receiving Long-term Antiretroviral Therapy. J Infect Dis. 2016 Feb 15;213(4):556-60. doi: 10.1093/infdis/jiv433. Epub 2015 Sep 2. PMID 26333941
- [Derived] Lee AJ, Bosch RJ, Evans SR, Wu K, Harrison T, Grant P, Clifford DB. Patterns of peripheral neuropathy in ART-naive patients initiating modern ART regimen. J Neurovirol. 2015 Apr;21(2):210-8. doi: 10.1007/s13365-015-0327-1. Epub 2015 Feb 13. PMID 25678143
- [Derived] Besson GJ, Lalama CM, Bosch RJ, Gandhi RT, Bedison MA, Aga E, Riddler SA, McMahon DK, Hong F, Mellors JW. HIV-1 DNA decay dynamics in blood during more than a decade of suppressive antiretroviral therapy. Clin Infect Dis. 2014 Nov 1;59(9):1312-21. doi: 10.1093/cid/ciu585. Epub 2014 Jul 29. PMID 25073894
- [Derived] Tenorio AR, Zheng Y, Bosch RJ, Krishnan S, Rodriguez B, Hunt PW, Plants J, Seth A, Wilson CC, Deeks SG, Lederman MM, Landay AL. Soluble markers of inflammation and coagulation but not T-cell activation predict non-AIDS-defining morbid events during suppressive antiretroviral treatment. J Infect Dis. 2014 Oct 15;210(8):1248-59. doi: 10.1093/infdis/jiu254. Epub 2014 May 1. PMID 24795473
- [Derived] Cillo AR, Krishnan S, McMahon DK, Mitsuyasu RT, Para MF, Mellors JW. Impact of chemotherapy for HIV-1 related lymphoma on residual viremia and cellular HIV-1 DNA in patients on suppressive antiretroviral therapy. PLoS One. 2014 Mar 17;9(3):e92118. doi: 10.1371/journal.pone.0092118. eCollection 2014. PMID 24638072
- [Derived] Lok JJ, Hunt PW, Collier AC, Benson CA, Witt MD, Luque AE, Deeks SG, Bosch RJ. The impact of age on the prognostic capacity of CD8+ T-cell activation during suppressive antiretroviral therapy. AIDS. 2013 Aug 24;27(13):2101-10. doi: 10.1097/QAD.0b013e32836191b1. PMID 24326304
- [Derived] Atkinson BE, Krishnan S, Cox G, Hulgan T, Collier AC. Anthropometric differences between HIV-infected individuals prior to antiretroviral treatment and the general population from 1998-2007: the AIDS Clinical Trials Group Longitudinal Linked Randomized Trials (ALLRT) cohort and NHANES. PLoS One. 2013 Jun 3;8(6):e65306. doi: 10.1371/journal.pone.0065306. Print 2013. PMID 23755215
- [Derived] Lok JJ, Bosch RJ, Benson CA, Collier AC, Robbins GK, Shafer RW, Hughes MD; ALLRT team. Long-term increase in CD4+ T-cell counts during combination antiretroviral therapy for HIV-1 infection. AIDS. 2010 Jul 31;24(12):1867-76. doi: 10.1097/QAD.0b013e32833adbcf. PMID 20467286